CLINICAL TRIAL: NCT03164005
Title: The Effects of VEGF-B Signaling Pathway in Obesity and Metabolic Disease
Acronym: Obesity
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chen Lulu, Head of Endocrinology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: 2016CFA025
Record Dates: First submitted 2017-05-13; First posted 2017-05-23 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Metabolic Disease
Keywords: VEGF-B
MeSH Terms: conditions — Obesity; Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma，Peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: subjects without metabolic diseases
- Group 2: subjects with metabolic diseases

SUMMARY:
The investigators will enroll about 120 subjects from the hospital's healthcare center. The investigators will collect the basic informations, blood pressure, body mass index, fasting blood glucose and fasting blood lipids of each subject. The investigators will collect the blood samples and then test them for fasting insulin levels, VEGF-B levels, the gene promoter region methylation status and the genomic protein methylation levels of the VEGF-B gene of the cells，and finally do the statistical analysis.

DETAILED DESCRIPTION:
The investigators will enroll about 120 subjects from the hospital's healthcare center, and these 120 subjects will be divided into four groups: normal weight with or without metabolic diseases and obesity with or without metabolic diseases. Each group has 30 subjects. The investigators will collect the basic information(name, gender，age, medical history，family history, etc.), blood pressure, body mass index, fasting blood glucose and fasting blood lipids of each subject from the healthcare center. The investigators will collect the blood samples of each subject,separate the plasma and then test the fasting insulin, VEGF-B levels by ELISA. The investigators will separate the peripheral blood mononuclear cells from the blood, and then test the gene promoter region methylation status of the VEGF -B gene by PCR and the bisulfite-modified sequencing and test the genomic protein methylation level of the VEGF-B gene by chromatin immunoprecipitation assay(CHIP) and real-time quantitative PCR of the cells，and finally do the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* NA

Exclusion Criteria:

* subjects with active history insulin treatment; and female participant pregnant at the time of recruitment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects without metabolic diseases , subjects with metabolic diseases
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Fasting insulin and blood VEGF-B levels | 3 days
  To investigate the relationship between blood pressure, BMI, fasting blood glucose, fasting blood lipids and fasting insulin and blood VEGF-B levels.

SECONDARY OUTCOMES:
The methylation status of VEGF-B gene promoter region and VEGF-B genomic protein methylation level . | 7 days
  To investigate the relationship between the methylation status of VEGF-B gene promoter region and VEGF-B genomic protein methylation level and obesity and metabolic disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Lulu, Principal Investigator — Department of Endocrinology, Union Hospital,Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Endocrinology, Union Hospital,Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No